CLINICAL TRIAL: NCT03545126
Title: Human CNS Tau Kinetics in Tauopathies
Acronym: TANGLES
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Association of Frontotemporal Degeneration (Unknown); Tau Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: 201703052
Record Dates: First submitted 2018-03-12; First posted 2018-06-04 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Progressive Supranuclear Palsy (PSP); Corticobasal Degeneration (CBD); Frontotemporal Dementia (FTD MAPT Mutation)
Keywords: Tauopathies
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Frontotemporal Dementia; Tauopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Progressive Supranuclear Palsy (PSP): N=12 Age: 18 and older Recruited participants will be given 13C6 Leucine through intravenous infusion (4mg/kg/hr for 16hrs), and CSF will be collected five times over 120 days (on approximately days 1-4, 5-10, 11-20, 21-60 and 61-120) after labeling.
  Interventions: Other: 13C6 Leucine
- Corticobasal Degeneration (CBD): N=8 Age: 18 and older Recruited participants will be given 13C6 Leucine through intravenous infusion (4mg/kg/hr for 16hrs), and CSF will be collected five times over 120 days (on approximately days 1-4, 5-10, 11-20, 21-60 and 61-120) after labeling.
  Interventions: Other: 13C6 Leucine
- Frontotemporal Dementia: MAPT: N=12 Family members with or at-risk of tau mutations (e.g. P301L) Age: 18 and older Recruited participants will be given 13C6 Leucine through intravenous infusion (4mg/kg/hr for 16hrs), and CSF will be collected five times over 120 days (on approximately days 1-4, 5-10, 11-20, 21-60 and 61-120) after labeling.
  Interventions: Other: 13C6 Leucine

INTERVENTIONS:
Other: 13C6 Leucine — Recruited participants will be given 13C6-labeled leucine through intravenous infusion (4mg/kg/hr for 16hrs)

SUMMARY:
The goal of this study is to characterize tau kinetics and tau aggregation in the human CNS and to test the hypothesis that tau kinetics are altered (i.e. increased production, decreased clearance, and increased aggregation rate) in tauopathies.

DETAILED DESCRIPTION:
Tauopathies are neurodegenerative diseases with tau pathology. These tauopathies are the most common pathology in neurodegenerative diseases, and they are reaching epidemic proportions. The rates of tau kinetics are central to understanding normal and abnormal processing and production and clearance of tau kinetics in humans to help understand the causes of tauopathy and evaluate tau-targeted therapeutics.

This study will utilize the Stable Isotope Labeling Kinetics (SILK) method to elucidate tau kinetics in vivo in the human central nervous system (CNS) and its alteration in tauopathies. A total of ~34 participants from 3 different neurodegenerative diseases: Frontotemporal Dementia (FTD), Corticobasal Degeneration (CBD), and Progressive Supranuclear Palsy (PSP), will be invited to enroll in the study.

Participants will be labeled with stable isotopes via 16hr intravenous infusion and CSF samples collected during subsequent lumbar puncture visits over ~120 days. CSF will be analyzed over time for the quantitation of labeled tau.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PSP, CBD, or FTD MAPT

Exclusion Criteria:

* Clotting disorder
* Active anticoagulation therapy
* Active infection
* Meningitis
* Recent syncope
* Current experimental treatment targeting Aβ or medications thought to influence Aβ production or clearance rates (benzodiazepines, muscarinic agents, or anti-epileptics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Progressive Supranuclear Palsy (PSP): N=12
  Corticobasal Degeneration (CBD): N=8
  Frontotemporal Dementia (FTD): MAPT: Family members with or at-risk of tau mutations (e.g. P301L) N=12
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Tau Fractional Turnover Rate (FTR) | 6 months
  Calculated by using CSF tau labeling and plasma free leucine.

SECONDARY OUTCOMES:
CSF Tau Absolute Concentration | 6 months
  Measured using labeled and unlabeled tau protein isoforms that will be immunoprecipitated and analyzed by mass spectrometry.
Tau Production Rate | 6 months
  Measured by FTR multiplied by CSF tau concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Bateman, MD, Principal Investigator — Washington University in Saint Louis Medical School; Nupur Ghoshal, MD, PhD, Principal Investigator — Washington University in Saint Louis Medical School
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time.